CLINICAL TRIAL: NCT01224327
Title: The Safety and Efficacy of Umbilical Cord Mesenchymal Stem Cells Infusion Via Hepatic Artery in Cirrhosis Patients.
Brief Title: Umbilical Cord Mesenchymal Stem Cells Infusion Via Hepatic Artery in Cirrhosis Patients
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Qingdao University (Other)
Responsible Party: Wang, Yangang MD, Stem Cell Research Center of Medical School Hospital of Qingdao University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MSCHC005
Record Dates: First submitted 2010-10-18; First posted 2010-10-20 (Estimated); Last update posted 2010-10-20 (Estimated); Status verified 2010-09

CONDITIONS: Liver Cirrhosis; Radiology; Mesenchymal Stem Cells; Umbilical Cord
Keywords: Liver cirrhosis; Radiology; Mesenchymal Stem Cells; Umbilical Cord
MeSH Terms: conditions — Liver Cirrhosis | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- umbilical cord mesenchymal stem cells (Experimental): Umbilical cord mesenchymal stem cells were infused to patients using interventional method via hepatic artery. After the catheter placed at proper hepatic artery was confirmed by angiography,umbilical cord MSCs were infused slowly for 15-20minutes.
  Interventions: Biological: umbilical cord Mesenchymal Stem Cells
- Conserved therapy (Active Comparator): Patients received comprehensive treatment including antiviral drugs, lowering aminotransferase and jaundice medicine.
  Interventions: Drug: Conserved therapy

INTERVENTIONS:
Biological: umbilical cord Mesenchymal Stem Cells — Umbilical cord mesenchymal stem cells were infused to patients using interventional method via hepatic artery. After the catheter placed at proper hepatic artery was confirmed by angiography,umbilical cord MSCs were infused slowly for 15-20minutes.
  Other Names: Mesenchymal Stem Cells
  Arms: umbilical cord mesenchymal stem cells
Drug: Conserved therapy — Oral or intravenous administration
  Other Names: Drug therapy
  Arms: Conserved therapy

SUMMARY:
The purpose of this study is to investigate the efficacy of umbilical cord mesenchymal stem cells (MSCs) infusion via hepatic artery in the treatment of liver cirrhosis.

DETAILED DESCRIPTION:
To investigate the efficacy of umbilical cord mesenchymal stem cells (MSCs) infusion via hepatic artery in the treatment of liver cirrhosis. Patients with liver cirrhosis were randomly separated into two groups. Umbilical cord MSCs were infused to patients using interventional method via hepatic artery for One group. After the catheter placed at proper hepatic artery was confirmed by angiography, umbilical cord MSCs were infused slowly for 15-20minutes. The control group accepted conserved therapy.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18~70 years.
* Liver cirrhosis
* written consent

Exclusion Criteria:

* The end-stage of liver cirrhosis.
* Severe problems in other vital organs(e.g.the heart,renal or lungs).
* Hepatocellular carcinoma or other malignancies
* Pregnancy
* sepsis
* Presence of significant extrahepatic biliary disease (e.g. CBD stone, PSC, etc.)
* Cardiac, renal or respiratory failure
* Active thrombosis of the portal or hepatic veins

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-10; Primary Completion 2012-10 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
The result of liver function and liver histological improvement. | every 4 weeks

SECONDARY OUTCOMES:
The disappearance or reduction of abdominal dropsy | every 4 weeks
The clinical symptom improve(including food appetite,debilitation,abdominal distension,edema of lower limbs ) | every 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Zibin Tian, MD, Study Director — The Affiliated Hospital of Qingdao University
Locations (1):
- Stem Cell Research Center of Medical School Hospital of Qingdao University, Qingdao, Shandong, China